CLINICAL TRIAL: NCT01647282
Title: Local Minocycline to Reduce Future Inflammation and Bone Loss in Periodontal Maintenance Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0314-12-FB
Record Dates: First submitted 2012-07-17; First posted 2012-07-23 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Moderate to Advanced Chronic Periodontitis
MeSH Terms: interventions — Minocycline; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sc/RP with minocycline micropheres (Experimental): Sc/RP is the subgingival mechanical removal of calculus and diseased cementum from the tooth root. Local application of minocycline microspheres will be done after scaling and root planing (Sc/RP) has been completed
  Interventions: Drug: locally-applied minocycline HCl (1 mg); Procedure: scaling and root planing (Sc/RP)
- Sc/RP alone (Active Comparator): Sc/RP is the subgingival mechanical removal of calculus and diseased cementum from the tooth root
  Interventions: Procedure: scaling and root planing (Sc/RP)

INTERVENTIONS:
Drug: locally-applied minocycline HCl (1 mg)
  Other Names: Arestin (minocycline microspheres) 1 mg
  Arms: Sc/RP with minocycline micropheres
Procedure: scaling and root planing (Sc/RP)

SUMMARY:
The purpose of this study is to determine the effect of local application of minocycline microspheres on the periodontal inflammation and bone loss prevention in patients diagnosed with moderate-severe chronic periodontitis within a periodontal maintenance program.

DETAILED DESCRIPTION:
The over-arching goal of this application is to initiate a program to involve undergraduate dental students and their patients in clinical research to evaluate the efficacy of dental therapy. Specifically, the purpose of this study is to determine the effect of local application of minocycline microspheres on the periodontal inflammation and bone loss prevention in patients diagnosed with moderate-severe chronic periodontitis on periodontal maintenance in the undergraduate clinic. Few studies evaluating locally-applied minocycline during periodontal maintenance therapy have been reported even though the drug is commonly used in this protocol. A 6-month treatment study by Meinberg et al. (2002), demonstrated that in moderate-to-advanced chronic periodontitis patients, scaling and root planing with subgingival minocycline resulted in improved pocket depths and less frequent bone height loss over one year than conventional periodontal maintenance. The prevention of bone loss and inflammation is key to maintaining teeth in function and comfort for the patient's lifetime. Patients from the UNMC College of Dentistry (and eventually Creighton University School of Dentistry) undergraduate periodontal clinic, who are already enrolled in periodontal maintenance therapy, will be recruited to participate in this study. The selected patients will continue their periodontal maintenance care but will be placed into either the test group (receiving minocycline in a periodontally inflamed pocket along with subgingival mechanical debridement) or the control group (receiving subgingival mechanical debridement alone). Radiographs will be taken at baseline and at the study's completion (24 months) to obtain bone loss data, and periodontal measurements and gingival crevicular fluid (GCF) will be used to monitor markers of inflammation and bone resorption. The hypothesis to be tested in this clinical trial is that the use of minocycline at baseline and 6 month intervals in conjunction with subgingival mechanical debridement will reduce interproximal bone height loss and periodontal inflammation more than mechanical debridement alone.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate-severe chronic periodontitis
* attending regular periodontal maintenance visits at UNMC COD
* one quadrant with at least one > 5 mm interproximal pocket and 3 posterior teeth

Exclusion Criteria:

* systemic diseases which impact periodontal inflammation and bone turnover
* drugs which significantly impact periodontal inflammation and bone turnover
* surgical periodontal therapy within the last year
* pregnant or breast-feeding females

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-10-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy C Killeen, DDS, MS, Principal Investigator — UNMC College of Dentistry
Locations (2):
- United States (2):
  - University of Nebraska, College of Dentistry, Lincoln, Nebraska
  - Creighton University School of Dentistry, Omaha, Nebraska

RESULTS

PARTICIPANT FLOW:
Groups:
- Sc/RP With Minocycline Micropheres: Sc/RP is the subgingival mechanical removal of calculus and diseased cementum from the tooth root. Local application of minocycline microspheres will be done after scaling and root planing (Sc/RP) has been completed
  locally-applied minocycline HCl (1 mg)
  scaling and root planing (Sc/RP)
- Sc/RP Alone: Sc/RP is the subgingival mechanical removal of calculus and diseased cementum from the tooth root
  scaling and root planing (Sc/RP)
Period: Overall Study
Arm/Group | Sc/RP With Minocycline Micropheres | Sc/RP Alone
Started | 30 | 30
Completed | 23 | 25
Not Completed | 7 | 5
Not completed — Physician Decision | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sc/RP With Minocycline Micropheres | Sc/RP Alone | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.3 (10.5) | 66.8 (12.1) | 67.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 14 | 16 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Interproximal Bone Height Loss, Probing Depth and Clinical Attachment Level Over 24 Months
Description: Changes in interproximal bone height loss were measured over the course of 24 months in two groups; patients receiving scaling and root planing alone in a deep periodontal pocket and those receiving scaling and root planing as well as minocycline microspheres in a deep periodontal pocket. These changes in interproximal bone height loss (mm) were determined via bitewing radiographs taken at baseline and 24 months and measured as distance from the cemento-enamel junction to the alveolar bone. Changes in probing depth (mm) were measured from the gingival margin to the depth of periodontal pocket. Changes in clinical attachment level (mm) were determined by adding the measure of gingival recession and the probing depth.
Time Frame: 24 months
Population: Patients included had moderate-severe chronic periodontitis with a >/= 5 mm interproximal, posterior pocket that bled upon probing. Participating patients had a history of regular periodontal maintenance therapy and no systemic disease (rheumatoid arthritis, osteoporosis, tetracycline allergy) or medications with bone-turnover significance.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Sc/RP With Minocycline Micropheres | Sc/RP Alone
Number analyzed (Participants) | 23 | 25
mm
  Interproximal Bone Loss Baseline | 3.78 (1.43) | 3.87 (1.11)
  Interproximal Bone Loss 24 Months | 3.57 (1.45) | 3.8 (1.13)
  Probing Depth - Baseline | 5.29 (0.62) | 5.48 (0.75)
  Probing Depth - 24 Months | 4.14 (0.89) | 3.96 (0.73)
  Clinical Attachment Level - Baseline | 5.42 (0.65) | 4.36 (1.05)
  Clinical Attachment Level - 24 Months | 5.81 (0.92) | 4.24 (0.66)

2. Secondary Outcome: Inflammatory Biomarkers Found in Gingival Crevicular Fluid: IL-1.
Description: The gingival crevicular fluid is analyzed biochemically and the levels of inflammatory biomarkers can be determined. Specific biomarkers are inherent in periodontal disease and have been shown to be indicative of periodontal breakdown within a pocket. In this study, the biomarker, IL-1 were assessed for their presence and quantity within the GCF samples taken from the experimental periodontal pockets at baseline and 24 months.
Time Frame: 24 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms/mL
Arm/Group | Sc/RP With Minocycline Micropheres | Sc/RP Alone
Number analyzed (Participants) | 23 | 25
picograms/mL
  Gingival Crevicular Fluid - Baseline | 9.29 (2.12) | 9.95 (1.98)
  Gingival Crevicular Fluid - 24 months | 10.30 (2.21) | 10.53 (2.16)

ADVERSE EVENTS:
Arm/Group | Sc/RP With Minocycline Micropheres | Sc/RP Alone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes